CLINICAL TRIAL: NCT05383157
Title: Brief Mindfulness Intervention for Chronic Pain in Ukraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Vinnitsa National Medical University (Other)
Responsible Party: Principal Investigator, Eric Garland, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0122U002551
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief mindfulness (Experimental): A 15-minute mindfulness intervention integrating mindful breathing and mindfulness of pain techniques.
  Interventions: Behavioral: Brief mindfulness; Other: Usual care
- Usual care (Active Comparator): 15 minutes of usual chronic pain care delivered in an academic pain clinic environment.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Brief mindfulness — Training in mindfulness focused on breathing and pain sensations to enhance decentering, meta-awareness, and interoceptive awareness.
  Arms: Brief mindfulness
Other: Usual care — Usual pain care as delivered in the clinic involving pain assessment and prescription of analgesics.

SUMMARY:
This is a pragmatic randomized controlled trial comparing a single 15-minute mindfulness-based intervention to usual care for patients with chronic pain in Ukraine being seen in a pain clinic.

ELIGIBILITY:
Inclusion Criteria:

* Physician-confirmed chronic pain-related diagnosis

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Other unstable illness judged by medical staff to interfere with study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Change from baseline to 20 minutes later.
  Single numeric rating scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.

SECONDARY OUTCOMES:
Pain unpleasantness | Change from baseline to 20 minutes later.
  Single numeric rating scale ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.
Positive affect | Change from baseline to 20 minutes later.
  Single numeric rating scale ranging from 0-10, with 0 indicating no positive affect and 10 representing very high levels of positive affect.
Desire for analgesic medication | Change from baseline to 20 minutes later.
  Single numeric rating scale ranging from 0-10, with 0 indicating no medication desire and 10 representing very high levels of medication desire.
Anxiety | Change from baseline to 20 minutes later.
  Single numeric rating scale ranging from 0-10, with 0 indicating no anxiety and 10 representing very high levels of anxiety.
Depression | Change from baseline to 20 minutes later.
  Single numeric rating scale ranging from 0-10, with 0 indicating no depression and 10 representing very high levels of depression.

OTHER OUTCOMES:
Decentering | Change from baseline to 20 minutes later.
  Three items from the The Metacognitive Processes of Decentering Scale rated on a numeric rating scale ranging from 0-10, with 0 indicating no decentering and 10 representing very high levels of decentering.
Self-transcendence | Change from baseline to 20 minutes later.
  Three items from the Nondual Awareness Dimensional Assessment rated on a numeric rating scale ranging from 0-10, with 0 indicating no transcendence and 10 representing very high levels of transcendence.

CONTACTS AND LOCATIONS:
Locations (1):
- Vinnitsa National Medical University, Vinnitsa, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided